CLINICAL TRIAL: NCT01145859
Title: Single-dose Pilot Study of Oral Rivaroxaban in Pediatric Subjects With Venous Thromboembolism
Brief Title: Rivaroxaban Pharmacokinetics/Pharmacodynamics (PK/PD) Study in Pediatric Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 12892; 2009-017313-30 (EudraCT Number)
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Venous Thrombosis; Pediatrics
Keywords: Venous Thrombosis; Pediatrics
MeSH Terms: conditions — Venous Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Weight adjusted dose with equivalent exposure compared to 10 mg or 20 mg doses in adults

SUMMARY:
The first study with rivaroxaban in pediatric subjects is a Phase I study, where the pharmacokinetic/pharmacodynamic (PK/PD) profile of rivaroxaban will be investigated to confirm that the exposure is comparable to adults. This study is a single dose study with multiple PK/PD measurements in pediatric subjects at the end of their Venous Thromboembolism (VTE) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects > 6 months and < 18 years of age at the time of administration of study drug.
* Patients who have completed treatment of VTE, but are considered to have risk for recurrence of VTE

Exclusion Criteria:

* Any major or clinically relevant bleeding during prior VTE treatment
* Abnormal coagulation tests within 7 days prior to study drug administration
* Severe renal impairment
* Planned invasive procedures prior to or after 24 hours of study drug administration

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2010-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters (AUC and Cmax) | From Day 1 to Day 2
Pharmacodynamics parameters (PT, aPTT and anti-factor Xa) | From Day 1 to Day 2

SECONDARY OUTCOMES:
Safety and tolerability of rivaroxaban in pediatric subjects | Day 1, day 2 plus 7 days follow up

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (34):
- United States (14):
  - Little Rock, Arkansas
  - Los Angeles, California
  - Orange, California
  - Gainesville, Florida
  - St. Petersburg, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Detroit, Michigan
  - New Hyde Park, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
- Australia (2):
  - Brisbane, Queensland
  - Parkville, Victoria
- Austria (2):
  - Vienna, Vienna
  - Linz
- Canada (3):
  - Edmonton, Alberta
  - Hamilton, Ontario
  - Toronto, Ontario
- France (4):
  - Clermont-Ferrand
  - Montpellier
  - Paris
  - Toulouse
- Lübeck, Schleswig-Holstein, Germany
- Crumlin, Dublin, Ireland
- Israel (2):
  - Jerusalem
  - Tel Litwinsky
- Italy (4):
  - Genova
  - Milan
  - Pavia
  - Torino
- Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Willmann S, Thelen K, Kubitza D, Lensing AWA, Frede M, Coboeken K, Stampfuss J, Burghaus R, Muck W, Lippert J. Pharmacokinetics of rivaroxaban in children using physiologically based and population pharmacokinetic modelling: an EINSTEIN-Jr phase I study. Thromb J. 2018 Dec 4;16:32. doi: 10.1186/s12959-018-0185-1. eCollection 2018. PMID 30534008
- [Derived] Kubitza D, Willmann S, Becka M, Thelen K, Young G, Brandao LR, Monagle P, Male C, Chan A, Kennet G, Martinelli I, Saracco P, Lensing AWA. Exploratory evaluation of pharmacodynamics, pharmacokinetics and safety of rivaroxaban in children and adolescents: an EINSTEIN-Jr phase I study. Thromb J. 2018 Dec 4;16:31. doi: 10.1186/s12959-018-0186-0. eCollection 2018. PMID 30534007
- [Derived] Willmann S, Becker C, Burghaus R, Coboeken K, Edginton A, Lippert J, Siegmund HU, Thelen K, Muck W. Development of a paediatric population-based model of the pharmacokinetics of rivaroxaban. Clin Pharmacokinet. 2014 Jan;53(1):89-102. doi: 10.1007/s40262-013-0090-5. PMID 23912563